CLINICAL TRIAL: NCT06882382
Title: Effects of Early Mobilization With Virtual Reality on Postoperative Respiratory Function, Exercise Capacity, and Pain in Children: A Randomized Controlled Trial
Brief Title: Use of Virtual Reality in Children Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Sabiha Bezgin, Mustafa Kemal University, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKU-SB-1
Record Dates: First submitted 2025-03-06; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Child, Only
Keywords: child; General Surgery; virtual reality

STUDY DESIGN:
Intervention Model Description: One group received virtual reality and physiotherapy, while the other group received only physiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): Only conventional physiotherapy was applied to this group, including normal joint movements, chest physiotherapy, and mobilization for 40 min each,
  Interventions: Other: conventional physiotherapy
- virtual reality group (Experimental): The CG received conventional physiotherapy, including normal joint movements, chest physiotherapy, and mobilization for 40 min each, whereas the other group received 20 min of VR application every day in addition to conventional physiotherapy interventions.
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: conventional physiotherapy — normal joint movements, chest physiotherapy, and mobilization for 40 min
  Arms: control group
Other: Virtual reality — normal joint movements, chest physiotherapy, and mobilization for 40 min and 20 min virtual reality
  Arms: virtual reality group

SUMMARY:
Aim: Early mobilization and exercise after surgery are very important to reduce the impact on lung function. The aim of this study was to compare the effects of early mobilization with virtual reality and conservative physiotherapy methods on pulmonary function, dyspnea, exercise capacity, pain, and kinesiophobia in children undergoing surgery.

Methods: The study included 27 children aged 5-18 years who underwent surgery. Among the children randomly divided into two groups, the control group (n = 14) received physiotherapy for 40 min twice a day for 3 days in the hospital after surgery, and the children were mobilized in and out of bed. In the virtual reality group (n = 13), in addition to physiotherapy practices, children were allowed to play virtual reality games for 20 min twice a day. Respiratory function, exercise capacity, and pain assessment were performed before surgery and before discharge.

DETAILED DESCRIPTION:
Aim: Early mobilization and exercise after surgery are very important to reduce the impact on lung function. The aim of this study was to compare the effects of early mobilization with virtual reality and conservative physiotherapy methods on pulmonary function, dyspnea, exercise capacity, pain, and kinesiophobia in children undergoing surgery.

Methods: The study included 27 children aged 5-18 years who underwent surgery. Among the children randomly divided into two groups, the control group (n = 14) received physiotherapy for 40 min twice a day for 3 days in the hospital after surgery, and the children were mobilized in and out of bed. In the virtual reality group (n = 13), in addition to physiotherapy practices, children were allowed to play virtual reality games for 20 min twice a day. Respiratory function, exercise capacity, and pain assessment were performed before surgery and before discharge.

ELIGIBILITY:
Inclusion criteria Between the ages of 5 and 18 undergone surgery for inguinal hernia, undescended testicle, hydrocele, cord cyst, umbilical hernia, circumcision, and distal hypospadias

Exclusion criteria

Children have visual and auditory sensory problems who required immobilization after surgery and had a chronic disease that would affect pulmonary function

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), ratio of forced expiratory volume in the first second to FVC (FEV1/FVC), peak expiratory flow rate (PEF), and forced mid-expiratory flow rate (FEF 25-75%) | 4 days
  The pulmonary function test was measured using a portable spirometer. According to American Torasic Society/European Respiratory Society (ATS/ERS) criteria, forced vital capacity (FVC), forced expiratory volume in the first second (FEV1), ratio of forced expiratory volume in the first second to FVC (FEV1/FVC), peak expiratory flow rate (PEF), and forced mid-expiratory flow rate (FEF 25-75%) were measured. The test was performed in the sitting position. The best of at least three technically acceptable manoeuvres with 95% agreement with each other was selected for statistical analysis.

SECONDARY OUTCOMES:
Respiratory muscle strength Assessment | 4 days
  Respiratory muscle strength was evaluated using an intraoral pressure measuring device. Maximal inspiratory pressure (MIP), inspiratory muscle strength, maximal expiratory pressure (MEP), and expiratory muscle strength were evaluated. MIP was measured using the intraoral pressure measurement method by performing rapid and deep inspiration in the residual volume after maximal expiration. MEP was recorded by performing rapid and deep expiration at total lung capacity after maximum inspiration. Children were verbally encouraged to record the best performance
Modified Borg Scale | 4 days
  Dyspnea evaluation was performed via the Modified Borg Scale (MBS). The scale, which was developed to measure the effort expended during physical exercise, consists of 10 items describing the severity of dyspnea according to its degree. According to the scale, it shows that the severity of dyspnea increases from 0 to 10
The 1-min step | 4 days
  The 1-min step (1-ST) test was performed. In the 1-ST, children were instructed to step reciprocally up and down a 6-in-high step for 1 min, and the number of steps taken was recorded.
Timed Up and Go Test | 4 days
  Participants were evaluated using the Timed Up and Go Test (TUG). The TUG is a clinical test that measures various components, including walking speed, postural control, functional mobility, and balance. The child was asked to get up from a chair without armrests, return to a sign 3 m away, and sit down. The duration was recorded in seconds
Numerical Pain Scale | 4 days
  The Numerical Pain Scale was used for pain assessment. The numerical pain scale assesses numerical values between 0 and 10 points
Kinesiophobia | 4 days
  The Tampa Scale of Kinesiophobia was used to assess kinesiophobia. The scale consists of 17 questions questioning the person's fear of movement and is calculated on a total score between 17 and 68. A high score on the scale indicates a high level of kinesiophobia
BMI | measured once, independent of time
  Height was measured and recorded in meters. Body weight was measured and recorded in kilograms. BMI was calculated by dividing body weight by height squared.
10 MWT test | 4 days
  In the 10 MWT, children walked at a normal walking speed within a 10-m section of a 14-m walking distance to prevent the effect of acceleration and deceleration phases of walking, and the time was recorded in seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Sabiha Bezgin, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bezgin S, Huzmeli I, Katayifci N, Yildirim BA, Atici A. Use of virtual reality in children undergoing surgery. Front Pediatr. 2025 Jul 16;13:1633310. doi: 10.3389/fped.2025.1633310. eCollection 2025. PMID 40740824